CLINICAL TRIAL: NCT00172094
Title: A Phase 2 Safety and Efficacy Study of NPS 1776 for the Acute Treatment of Migraine Headaches
Brief Title: Safety and Efficacy of NPS 1776 in the Acute Treatment of Migraine Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL1776-005
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Migraine Headache
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): PLACEBO
  Interventions: Drug: PLACEBO
- 2 (Experimental): 400 mg 1776 powder
  Interventions: Drug: NPS 1776 (400 mg)
- 3 (Experimental): 1776 (800 mg)
  Interventions: Drug: NPS 1776 (800 mg)

INTERVENTIONS:
Drug: NPS 1776 (800 mg) — NPS 1776 (800 mg) powder
  Other Names: NPS 1776
  Arms: 3
Drug: PLACEBO — Placebo in non-carbonated fruit flavored drink (150 ml)
  Arms: 1
Drug: NPS 1776 (400 mg) — NPS1776 in powdered form to be mixed with a non-carbonated fruit flavored drink
  Other Names: NPS1776
  Arms: 2

SUMMARY:
The purpose of this study was to evaluate the effectiveness and safety of a single oral dose of NPS 1776 in the acute treatment of migraine pain and associated symptoms.

DETAILED DESCRIPTION:
Migraine, the most common cause of recurrent severe or disabling headache, is diagnosed on the basis of a clinical history of intermittent headache with autonomic, constitutional, and neurologic disturbances.

Many antiepileptic drugs (AEDs) have demonstrated efficacy as acute and/or prophylaxis therapy for migraine, even though the mechanism of action of the various AEDs is poorly understood.

NPS 1776, isovaleramide, is a neutral aliphatic amide. The mechanism by which NPS 1776 exerts its therapeutic actions in nonclinical animal models of disease is unclear. The same is true for many antiepileptics on the market today. NPS 1776 does not appear to bind directly to various CNS receptor centers, although it shows a broad range of anticonvulsant activity in multiple animal models of seizures. This broad profile of anticonvulsant activity is similar to that of valproic acid (VPA), and may also predict NPS 1776 efficacy in the treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of migraine for at least a year prior to screening.
2. Experiences 2-10 migraine headaches per month (with at least 24 hours between episodes) and no more than 15 headache days per month in the 3 months prior to screening.
3. Ability and willingness to arrive at the investigator's center within 1 hour (±5 min) of migraine pain onset (defined as pain that is consistent with the subject's usual migraine and is of at least moderate severity).
4. Ability and willingness to abstain from taking medications not allowed by the protocol and to meet phone and check-in criteria.
5. Ability and willingness to undergo a comprehensive urine toxicology screen for both licit and illicit drugs.
6. Ability and willingness to complete a migraine-history diary from screening to treatment with study drug and a migraine-treatment diary from discharge through the remainder of the 24-hour period following study-drug treatment.

Exclusion Criteria:

1. Unstable or uncontrolled significant metabolic, hepatic, renal, hematological, pulmonary, gastrointestinal, urological, neurological (except migraine headaches), or psychiatric disorders.
2. Severe or acute cardiovascular or cerebrovascular disease, uncontrolled hypertension, or basilar or hemiplegic migraines.
3. History of hypersensitivity, allergies, or nonresponse to valproic acid.
4. Have taken VPA or other AED in the 30 days prior to screening, or are taking a migraine prophylaxis treatment other than a stable dose of propranolol or tricyclic antidepressant.
5. Migraine attacks that in the investigator's opinion are associated with intractable nausea and/or vomiting.
6. Any acute or chronic condition that in the investigator's opinion would limit the subject's ability to complete and/or participate in this clinical study or would place the subject at increased risk.
7. Have newly started or changed the dose of either feverfew or magnesium (above 200 mg, the amount in common daily supplements) within 3 months prior to screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2003-12-31 (Actual); Primary Completion 2004-06-30 (Actual); Study Completion 2004-07-31 (Actual)

PRIMARY OUTCOMES:
The response rate at 2 hours post-dose such that the percentage of subjects whose migraine pain-intensity score is none [0] or mild [1] at 2 hours post-dose, after a baseline pain intensity of moderate [2] or severe [3] | 2 hours post-dose

SECONDARY OUTCOMES:
Pain-free rate at 2 hours post-dose | 2 hours post-dose
Response rate up to 48 (±24) hours post-dose | 48 hours post-dose
Recurrence rate of migraine headache within 24 hours post dose | 24 hours post-dose
Time to recurrence of migraine within 24 hours post-dose | 24 hours post-dose
Area under the migraine pain curve in visual analogue scale (VAS) 0 4 hours post-dose | 4 hours post-dose
VAS pain reduction: peak pain reduction in VAS score 0-4 hours post-dose | 4 hours post-dose
Presence of nausea/vomiting, sensitivity to sound/light, skin sensitivity (cutaneous allodynia), intracranial sensitivity | 24 hours post-dose
Brush allodynia | 24 hours post-dose
Muscle tenderness | 24 hours post-dose
Functional disability | 24 hours post-dose
Use of rescue medication | 4 hours post-dose
Time to meaningful pain relief | 2 hours post-dose
Global Subject Impression (GSI) | 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (22):
- United States (22):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - North County Neurological Associates, Oceanside, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Clinical Innovations, Santa Ana, California
  - California Medical Clinic for Headache, Santa Monica, California
  - The New England Center for Headache, Stamford, Connecticut
  - University Clinical Research, Inc, Pembroke Pines, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - MedTrial Boston, Wellesley Hills, Massachusetts
  - Michigan Head-Pain & Neurological Institute, Ann Arbor, Michigan
  - Mercy Health Research, Chesterfield, Missouri
  - Headache Care Center/ Clinvest, Springfield, Missouri
  - University of Medicine and Dentistry, New Jersey School of Osteopathic Medicine, Moorestown, New Jersey
  - Neuroscience Center of Northern New Jersey, Morristown, New Jersey
  - Headache Wellness Center, Greensboro, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Neurology Ctr. of Ohio, Toledo, Ohio
  - The Neurology Clinic, Portland, Oregon
  - Thomas Jefferson University Hospital/ Jefferson Headache Center, Philadelphia, Pennsylvania
  - Houston Headache Clinic, Houston, Texas
  - Neurology & Neurosurgery Associates of Tacoma, Inc., PS, Tacoma, Washington

REFERENCES:
- See also: American Headache Society - Site dedicated to the study and treatment of headaches of all types including but not limited to migraines. — http://www.ahsnet.org